CLINICAL TRIAL: NCT05832294
Title: Finding a Biomarker for Acute Neuromodulation Effects in Adolescent Depression: A Pilot Study
Brief Title: Finding a Biomarker for Acute Neuromodulation Effects in Adolescent Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Giacobbe, Clinical Head, Associate Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5439
Record Dates: First submitted 2023-03-13; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Recruitment

STUDY DESIGN:
Intervention Model Description: Single-blinded sham-controlled between-subjects design with two arms.
Who Masked: Participant
Masking Description: Single-blinded sham-controlled between-subjects design with two arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Stimulation (Sham Comparator): 15 Depressed adolescents will undergo emotional processing tasks (within and outside the fMRI scanner) after one session of sham rTMS
  Interventions: Device: Sham rTMS
- Active Stimulation (Active Comparator): 15 Depressed adolescents will undergo emotional processing tasks (within and outside the fMRI scanner) after one session of active rTMS
  Interventions: Device: Treatment rTMS

INTERVENTIONS:
Device: Treatment rTMS — Depressed adolescents will undergo emotional processing tasks (within and outside the fMRI scanner) after one session of 1) sham rTMS (n = 15) or 2) active rTMS (n = 15). Prior to stimulation, expectancy for symptomatic benefit will be assessed with a standardized scale and a semi-structured interview conducted regarding their perception of rTMS. After the one-day randomized controlled phase, participants can then enter an open-label active rTMS treatment phase for 4 weeks. Eligible patients who decline the study and open-label treatment phase will be invited to participate in a semi-structured interview to explore their perceptions toward rTMS.
  Arms: Active Stimulation
Device: Sham rTMS — Depressed adolescents will undergo emotional processing tasks (within and outside the fMRI scanner) after one session of 1) sham rTMS (n = 15) or 2) active rTMS (n = 15). Prior to stimulation, expectancy for symptomatic benefit will be assessed with a standardized scale and a semi-structured interview conducted regarding their perception of rTMS. After the one-day randomized controlled phase, participants can then enter an open-label active rTMS treatment phase for 4 weeks. Eligible patients who decline the study and open-label treatment phase will be invited to participate in a semi-structured interview to explore their perceptions toward rTMS.
  Arms: Sham Stimulation

SUMMARY:
This pilot study aims to examine the feasibility of recruiting depressed adolescents to examine changes in emotional processing and in neural responses to emotional stimuli after one session of rTMS (which is followed by an open-label phase of 4 weeks active rTMS).

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a promising treatment for adolescent depression but clinical trials have been hampered by a lack of dose optimization studies and high placebo rates. While rTMS does not produce mood changes until after weeks of treatment, unconscious changes in emotional processing have been found even after one session of stimulation. It is unknown whether one session of rTMS produces changes in neural activity to emotional stimuli in depressed adolescents. If acute rTMS can reliably produce changes in neural activity associated with emotional processing it could be a biomarker to aid future dose-finding studies. A one-session protocol allows experimenters to truthfully reduce expectancy of mood change and reduce placebo effects. This study will examine the feasibility of recruitment and using a one-session protocol to find a biomarker for acute rTMS effects. A single-blinded sham-controlled design will be used. Depressed adolescents will undergo: 1) sham stimulation (n=15) or 2) active stimulation with intermittent theta burst stimulation (iTBS) (n=15) for one session prior to assessment of brain activity in response to emotional stimuli in a fMRI and other emotional processing tasks. This one day randomized controlled phase can then lead into an open-label treatment phase active rTMS for 4 weeks. The primary outcome will be recruitment rates with a secondary outcome of estimating the magnitude of difference detectable in cortico-limbic activity between groups. This study assesses the feasibility of a novel paradigm to help improve clinical trials for neuromodulation in depressed adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients between ages 14-21
2. Diagnosis of major depressive disorder as defined by the Diagnostic and Statistical Manual fifth edition (DSM-5)
3. Hamilton Rating Scale for Depression (17-item) score of at least 20
4. At least one failed adequate antidepressant trial
5. On a stable antidepressant regimen for at least 4 weeks before treatment which can continue during treatment and agreement to not make changes or additions to psychotropic medications during the course of their participation in the study
6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, delusional disorder, post-traumatic stress disorder, obsessive compulsive disorder, autism spectrum disorder
2. Active neurologic disease
3. Any lifetime history of seizures
4. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
5. Current active suicidal ideation
6. Personality disorder deemed to be the primary pathology
7. Taking more than 2 mg lorazepam (or an equivalent) or any anticonvulsant
8. Previous rTMS treatment

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 2 years
  What is the sufficient time to recruit depressed adolescents from Sunnybrook Health Sciences Centre who provide informed consent for a study examining the effects of one-session rTMS on brain function as measured by fMRI

SECONDARY OUTCOMES:
estimating the magnitude of difference detectable in cortico-limbic activity between groups | 2 years
  How many sessions of rTMS is sufficient to produce changes in emotional processing and associated cortico-limbic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No